CLINICAL TRIAL: NCT06379633
Title: Virtual Reality Exposure for Socially Anxious Adolescents: A Randomized Controlled Trial (RCT)
Brief Title: Virtual Reality Exposure for Socially Anxious Adolescents
Acronym: VIRTUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Utrecht University (Other)
Responsible Party: Principal Investigator, Dirk Hermans, Full professor, PhD, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: s67010
Record Dates: First submitted 2024-04-02; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Social Anxiety
Keywords: virtual reality exposure; social anxiety; adolescents; inhibitory learning theory; predictors; youth; mental health; mechanisms
MeSH Terms: conditions — Psychological Well-Being | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the three conditions and will remain in that condition throughout the training sessions.
Who Masked: Outcomes Assessor
Masking Description: All pre-assessments and post-assessment will be conducted by researchers who will be blind to the participants' allocated condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality exposure (VRE) (Experimental): Participants in the VRE condition will be exposed to various VR-based one-on-one and group social interactions which tend to elicit anxiety. That is, commonly feared situations and events (e.g., raising your hand in class, saying no to a friend, ordering food at a restaurant, calling a classmate to invite them to hang out) will be recreated in the virtual environments. Exercises will be tailored to the participant and provided by clinical psychologists under supervision of experienced CBT therapists (and supervisors). To deliver VRE we will utilize a dynamic and interactive VR-software called 'Social Worlds' developed by CleVR. It has various functions and capabilities (e.g., role-playing, walking around, change of perspective, alteration of dialogue style, number of avatars present in the virtual environment) which enables individualized exposure.
  Interventions: Behavioral: (Virtual reality) exposure
- In vivo exposure (IVE) (Active Comparator): Similarly to VRE, participants in the IVE condition will be exposed to various one-on-one and group social interactions which tend to elicit anxiety, but they will do so in real-life. The exposure exercises here also will be determined in consultation with the participant. Depending on the given exposure exercise, exposure will either take place at the training location or in its neighborhood (e.g., nearby supermarkets, subway stations, cafes, buses). Exercises will be tailored to the participant and provided by clinical psychologists under supervision of experienced CBT therapists (and supervisors). Importantly, participants will undergo the same amount of exposure sessions as in the VRE condition (to keep exposure time constant).
  Interventions: Behavioral: In vivo exposure
- Waitlist (No Intervention): The participants in the WL condition will complete the assessments at the same time points as in the active conditions but will not receive any of the sessions until post-assessment has been completed. Then they will be randomly assigned to one of the two active conditions (VRE or IVE).

INTERVENTIONS:
Behavioral: In vivo exposure — Exposure in vivo involves the confrontation with fear-evoking situations in real life.
  Arms: In vivo exposure (IVE)
Behavioral: (Virtual reality) exposure — Exposure in virtual reality involves the confrontation with fear-evoking situations which are generated by a computer using VR technology.
  Arms: Virtual reality exposure (VRE)

SUMMARY:
Overall in this project, the primary goal is to evaluate the efficacy of virtual reality exposure (VRE) for adolescents with elevated social anxiety using a three-arm randomized controlled trial: (1) virtual reality exposure (VRE); (2) in vivo exposure (IVE); and (3) waitlist (WL) - the control condition.

It is predicted that both VRE and IVE will be more successful in decreasing social anxiety symptoms than the WL condition at post-assessment and that VRE will be as effective as in vivo in reducing social anxiety symptoms. Furthermore, it is expected that there will be no difference between the two active conditions in the long term (at 3- months & 6-months follow up). Similar results are expected in the secondary outcome measures, intended to capture the participants' general well-being.

Moreover, the study has the following (secondary) objectives:

* To elucidate potential working mechanisms of VRE and IVE
* To identify predictors of adolescents' response to VRE and IVE
* To assess to what extent adolescents accept VRE and IVE and how they experience it

DETAILED DESCRIPTION:
This study is going to be a single-blinded, randomized controlled trial (RCT) with three arms: VRE, IVE, and a WL condition. It will follow a mixed-subjects design with condition as a between factor and measurement time-points as a within factor. Due to the study's goal to unravel the effects of VRE, the focus of the intervention will be on exposure in both active conditions (without explicitly including other treatment components like cognitive restructuring). The intervention will take place either at participants' schools or at KU Leuven (i.e., PraxisP - the outpatient treatment facility of the Faculty of Psychology and Educational Sciences, PSI - Psychological Institute) depending on the participants' preference and availability. In case this is not possible, neighboring healthcare practices will be explored as an alternative option. In any case, the training will be held in a separate, private room where the privacy of the participant can be guaranteed. Each active condition will comprise of 7 training sessions in total approximately 90 minutes each.

At pre-assessment, all primary and secondary outcome measures and most of the predictors will be assessed approximately one week prior to the first session. The outcome measures will be re-assessed during the post-assessment (one week after the last session) and the follow up assessments (3-months & 6-months following the post assessment). During the training sessions, measurements of the mechanisms, remaining predictors, and participant feedback will be acquired and at mid-assessment an additional measurement of the primary outcome measures (e.g., social anxiety measures) will be obtained. Moreover, a brief social anxiety measure will also be conducted on a weekly basis to record symptom-related changes from session to session. Following the training, a qualitative interview will be conducted. This semi-structured interview will be conducted in a convenience sample of participants from both active conditions (e.g., 10-16 participants per condition due to pragmatic considerations and based on general recommendations as to when theoretical data saturation can be reached) to investigate VRE's acceptability and to compare it to IVE. To decrease demand effects, the (online) interview will be conducted by an independent interviewer (e.g., not the therapist) and will be audio-taped so that the interviewer can focus solely on the interaction.

Moreover, in line with good clinical practice and individualized treatment, the specific nature and content of the exposure exercises will be determined for each participant individually by presenting them with an extensive list of the possible exercises (e.g., ordering food in a restaurant, asking a question in class, engaging in a group conversation) in combination with a functional analysis. To ensure that the active conditions are comparable, the IVE condition will be matched to the VRE condition in terms of exposure duration and homework assignments will not be actively encouraged in both conditions. The crucial difference between the two active conditions is that in the IVE condition the exercises take place in real life, whereas in VRE the exercises take place in virtual reality. For the WL condition, the (primary and secondary) outcome measures will be administered before, during, and after the given waiting period (i.e., duration of training sessions) at the same instances as with the active conditions. After that time, participants in the WL condition will have the opportunity to be randomized into IVE and VRE.

ELIGIBILITY:
Inclusion:

* Elevated levels of social anxiety (as per the Social Phobia Inventory; ≥ 19)
* Fluent in Dutch
* 12-16 years old

Exclusion

* Severe social anxiety disorder
* Severe depression
* Psychotic symptoms
* Severe suicidal thoughts and / or severe self-harm
* Severe substance use
* Benzodiazepine use and / or a change of psychoactive medication usage (dose, type)
* Autism spectrum disorder (ASD) diagnosis
* Current ongoing psychological treatment (or waitlisted) for anxiety disorders and or depression
* Other urgent psychopathologies and/or mismatch between participants' clinical presentation and the offered training
* Exposure therapy for social anxiety disorder in the past 2 years
* Another person from the same household is participating in the study
* Eligible for VR as per the following criteria:
* History of extreme/severe motion sickness (e.g., car sick, sea-sick) and / or experiencing extreme/severe symptoms of motion sickness during 3D movies
* Stereoscopic vision problem or a balance problem that would hinder the VR experience;
* History of seizures, seizure disorder or epilepsy

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Brief version of the Social Phobia and Anxiety Inventory (SPAI-18) | Pre-assessment, after 4 weeks, after 8 weeks, follow-up(after 20 weeks), follow up(after 32 weeks)* *Due to practical reasons (e.g., school vacation) the exact number of weeks may change. This applies for all the timepoints except pre-assessment.
  General measure of social anxiety
Liebowitz Social Anxiety Scale for Children and Adolescents (LSAS-CA) - Avoidance subscale | Pre-assessment, after 4 weeks, after 8 weeks, follow-up(after 20 weeks), follow up(after 32 weeks)*
  Avoidance measure of social anxiety
Behavioral assessment task (BAT) - Peak anxiety | Pre-assessment, after 8 weeks*
  Subjective units of distress (SUD) measured on a visual analogue scale (VAS); administered immediately after the BAT

SECONDARY OUTCOMES:
Brief Resilience Scale (BRS) | Pre-assessment, after 4 weeks, after 8 weeks, follow-up(after 20 weeks), follow up(after 32 weeks)*
  General measure of resilience
Multidimensional Adolescent Functioning Scale (MAFS) - Peer and General functioning subscales | Pre-assessment, after 4 weeks, after 8 weeks, follow-up(after 20 weeks), follow up(after 32 weeks)*
  General measure of psychosocial functioning
Revised Children's Anxiety and Depression Scale (RCADS) | Pre-assessment, after 4 weeks, after 8 weeks, follow-up(after 20 weeks), follow up(after 32 weeks)*
  General measure of depression and anxiety + Predictor
Self-Efficacy Questionnaire for Children (SEQ-C) - Social efficacy subscale | Pre-assessment, after 4 weeks, after 8 weeks, follow-up(after 20 weeks), follow up(after 32 weeks)*
  General measure of social self efficacy and mechanism
Social Phobia Weekly Summary Scale (SPWSS) | Pre-assessment, every training week (up to 7 weeks after pre-assessment), after 8 weeks, follow-up(after 20 weeks), follow up(after 32 weeks)*
  Weekly measure of social anxiety
Liebowitz Social Anxiety Scale for Children and Adolescents (LSAS-CA) - Fear subscale | Pre-assessment, after 4 weeks, after 8 weeks, follow-up(after 20 weeks), follow up(after 32 weeks)*
  Secondary measure of fear regarding specific social situations
Adolescent Social Cognitions Questionnaire (ASCQ) | Pre-assessment, after 8 weeks, follow-up(after 20 weeks), follow up(after 32 weeks)*
  Secondary outcome and mechanism & predictor
Behavioral assessment task (BAT) - Anticipatory anxiety | Pre-assessment, after 8 weeks*
  Subjective units of distress (SUD) measured on a visual analogue scale (VAS) immediately before the BAT
Behavioral assessment task (BAT) - Physiological assessment | Pre-assessment, after 8 weeks*
  Mean heart rate measured during the BAT
Behavioral assessment task (BAT) - Physiological assessment | Pre-assessment, after 8 weeks*
  Heart-rate variability measured during the BAT
Behavioral assessment task (BAT) - Physiological assessment | Pre-assessment, after 8 weeks*
  Skin conductance response measured during the BAT
Behavioral assessment task (BAT) - Task duration | Pre-assessment, after 8 weeks*
  Duration of task in seconds
Behavioral assessment task (BAT) - Confederate rating | Pre-assessment, after 8 weeks*
  During the BAT, the confederate will rate the participants' social anxiety and performance on a 5-point Likert scale

OTHER OUTCOMES:
Behavioral inhibition system / behavioral activation system scale (BIS/BAS) | Pre-assessment
  Predictor
Experiences in Close Relationship Scale - Relationship Structures (ECR-RS) | Pre-assessment
  Predictor
Immersive Tendency Questionnaire (ITQ) - Factor Involvement | Pre-assessment
  Predictor
Unified Theory of Acceptance and Use of Technology (UTAUT-A) - Attitudes subscale | Pre-assessment
  Predictor
Unified Theory of Acceptance and Use of Technology (UTAUT-EC) - Expectancy subscale | Pre-assessment
  Predictor
VR experience, motivation, need for connection/relatedness, openness to experiences | Pre-assessment
  Predictors - Each construct mentioned above will be measured on a single VAS
Preference for treatment question | Pre-assessment
  Predictor measured as a binary outcome
Credibility and Expectancy Questionnaire (CEQ) | 1 week after pre-assessment*
  Predictor
Working Alliance Inventory-Short Form (WAI-S) | 2 and 6 weeks after pre-assessment*
  Predictor
Exposure log questions - expectancy violation & expectancy change | Weekly training sessions (up to 7 weeks after pre-assessment)*
  Mechanism - Measures related to threat expectancies (e.g., likelihood of threat expectancy, how bad it would be if it occurred) and threat occurrence (e.g., extent to which it occurred, surprise, relief, adjusted threat expectancy).
  These variables will be collected prior to and after the exposure exercises and will be primarily assessed using visual analogue scales (VASs).
Exposure log open-ended questions - expectancy violation & expectancy change | Weekly training sessions (up to 7 weeks after pre-assessment)*
  Mechanism - open ended questions (e.g., what they learned, how they know that their threat expectancy did not occur) will also be asked to provide further context and to provide more insights into the participants' responses.
Exposure log questions - within- & between- session habituation | Weekly training sessions (up to 7 weeks after pre-assessment)*
  Mechanism - Subjective units of distress prior (anticipatory fear/anxiety) and after the exposure exercises (end fear/anxiety & peak fear/anxiety).
  They will be measured using visual analogue scales (VASs)
Exposure log question- Self-efficacy | Weekly training sessions (up to 7 weeks after pre-assessment)*
  Mechanism - Visual analogue scale (VAS) measuring self-efficacy regarding handling social situations
Exposure log question - Presence | Weekly training sessions (up to 7 weeks after pre-assessment)*
  Mechanism - Only in the VRE condition a measure of presence (e.g., measuring how present they feel in the VR environment) will be collected for each exposure exercise.
Exposure log questions - Participant feedback | Weekly training sessions (up to 7 weeks after pre-assessment)*
  During each training session, visual analogue scales (VASs) will be administered to measure exercise difficulty, exercise usefulness/relevance, use of safety behaviors, and motivation to participate in the next session
Acceptability interview | Between post-assessment and first follow-up (between 8 and 20 weeks after pre-assessment)
  A semi-structured interview will be conducted in a convenience sample of participants from both active conditions (e.g., 10 participants per condition) to investigate VRE's acceptability and to compare it to IVE.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Hermans, PhD, Principal Investigator — KU Leuven
Locations (1):
- Psychological Institute (PSI) of KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
There are no concrete plans to upload individual participant data on to any platforms. However, if other researchers request for the pseudo-anonymized data, then an agreement can be made to share the data.

REFERENCES:
- [Derived] Uduwa Vidanalage ES, De Lee J, Hermans D, Engelhard IM, Scheveneels S, Meyerbroker K. VIRTUS: virtual reality exposure training for adolescents with social anxiety - a randomized controlled trial. BMC Psychiatry. 2025 Apr 18;25(1):401. doi: 10.1186/s12888-025-06756-w. PMID 40251576